CLINICAL TRIAL: NCT04740879
Title: The Effects of the "Be Mindful" Intervention in Previously Depressed College Students Currently Experiencing Subclinical Symptoms of Depression
Brief Title: The Effects of the Be Mindful Intervention in Previously Depressed Individuals Experiencing Subclinical Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Meghan Bauer, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005212; SU-20-01 (Other Grant/Funding Number: State University of New York at Buffalo)
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms; Major Depressive Disorder, Recurrent, in Remission
Keywords: Mindfulness Based Cognitive Therapy; Be Mindful Intervention; Past Major Depressive Disorder; Major Depressive Disorder; Depressive Symptoms; Mechanisms of Change
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Intervention condition will be provided with access to the 4-week online Mindfulness-Based Cognitive Therapy course "Be Mindful" immediately after randomization to group.
  Interventions: Behavioral: Be Mindful
- Waitlist Control (Other): The Waitlist Control condition will be provided with access to the 4-week online Mindfulness-Based Cognitive Therapy course "Be Mindful" approximately 4 months after randomization to group.
  Interventions: Behavioral: Be Mindful

INTERVENTIONS:
Behavioral: Be Mindful — The online 4-week Be Mindful intervention was designed to follow the same outline as typical in-person 8-week MBCT courses. Week 1 and Week 2 introduce the topic of mindfulness and encourage its daily use, whereas Week 3 and Week 4 teach the individual to decenter from thoughts and utilize mindfulness when coping with stressors. Each week focuses on a separate mindfulness topic, which is initially presented to the individual in a short (under 5 minute) video containing didactic information and an overview of the experiential activities that will be introduced in subsequent videos. The intervention is provided entirely through audio, video, and text provided on the Be Mindful website (BeMindfulOnline.com).

SUMMARY:
This study is designed to help individuals cope with their current depressive symptoms by providing them access to a 4-week online Mindfulness-Based Cognitive Therapy: Be Mindful. Research has shown that completion of the Be Mindful intervention can reduce depressive symptoms in a community sample, and this study aims to evaluate if it can also help reduce depressive symptoms in individuals with a confirmed history of depression. Participants will either receive the intervention at the start of the study or four months after the start of the study (i.e., at 3-month follow-up), which will allow research staff to assess if reductions in depression are due to the intervention or something else. Research staff will also evaluate if the reduction in depressive symptoms lasts over the three months following intervention, and will investigate possible reasons for the change in depression (i.e., why the intervention produces change).

DETAILED DESCRIPTION:
Participant outcome variables will be assessed weekly for the first month after baseline. This will include the primary dependent variable (i.e., depressive symptoms), but will also include variables that will be explored as potential mechanisms of change (i.e., mindfulness, decentering, rumination, worry, self-compassion, and dysfunctional attitudes). The final weekly assessment will represent the Post-Intervention assessment.

Brief follow-up assessments of the primary dependent variable will be given 1-month and 2-months after the final weekly questionnaire. There will be a 3-month assessment that measures potential mechanisms of change in addition to the primary dependent variable.

After the 3-month follow-up, the Waitlist Control condition will be given access to the intervention. All participants (i.e., in both conditions) will be asked to complete another month of weekly questionnaires. These questionnaires will be identical to the first set of weekly questionnaires, and will allow mechanisms of change to be evaluated in the Waitlist Control condition.

ELIGIBILITY:
Inclusion Criteria:

* currently experiencing mild to moderate depressive symptoms (Patient Health Questionnaire 9 Current scores between 5 and 14)
* meet Diagnostic and Statistical Manual of Mental Disorders (fifth edition; DSM-5) criteria for Past Major Depressive Disorder (determined by clinical interview)

Exclusion Criteria:

* responses suggest they have never experienced a Major Depressive Episode
* responses suggest they are not currently experiencing sub-threshold symptoms of depression
* they state they are not open to learning mindfulness or meditation techniques
* they indicate they are currently receiving therapeutic treatment for depression or stress management elsewhere
* they indicate their age is not between 18 and 65
* they state they do not currently live in New York State

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mean Change in Depressive Symptoms from Baseline as Measured by the Patient Health Questionnaire 9 Post-Intervention | weekly during intervention, approximately 1-2 months
  Participants are asked to rate items on a scale of 0 (Not at all) to 3 (Nearly every day).
Mean Change in Depressive Symptoms from Baseline as Measured by the Patient Health Questionnaire 9 at 3-Month Follow-Up | at regular intervals until 3-month follow-up (approximately 4-5 months after the start of the study)
  Participants are asked to rate items on a scale of 0 (Not at all) to 3 (Nearly every day).

SECONDARY OUTCOMES:
Mean Change in Mindfulness from Baseline as Measured by the Five Factor Mindfulness Questionnaire Short Form | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 1 (never or rarely true) to 5 (very often or always true).
Mean Change in Decentering from Baseline as Measured by the Toronto Mindfulness Scale | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 0 (not at all) to 4 (very much).
Mean Change in Rumination from Baseline as Measured by the Ruminative Response Questionnaire | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 1 (Almost never) to 4 (Almost always).
Mean Change in Worry from Baseline as Measured by the Penn State Worry Questionnaire | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 1 (Not at all typical of me) to 5 (Very typical of me).
Mean Change in Self-Compassion from Baseline as Measured by the Self-Compassion Scale Short Form | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 1 (Almost never) to 4 (Almost always).
Mean Change in Dysfunctional Attitudes from Baseline as Measured by the Dysfunctional Attitudes Scale (Short Form 1) | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 1 (totally agree) to 4 (totally disagree).
Mean Change in Dysfunctional Attitudes from Baseline as Measured by the Rosenberg Self-Esteem Scale | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 0 (strongly disagree) to 3 (strongly agree).
Mean Change in Dysfunctional Attitudes from Baseline as Measured by the Single-Item Self-Esteem Scale | through study completion, which can take up to 6 months
  Participants are asked to rate items on a scale of 1 (Not Very True of Me) to 5 (Very True of Me).

CONTACTS AND LOCATIONS:
Overall Officials: Meghan E Bauer, MA, Principal Investigator — State University of New York at Buffalo; John E Roberts, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo (SUNY at Buffalo), Buffalo, New York, United States